CLINICAL TRIAL: NCT04282837
Title: Data-driven Clustering for Metabolic Classification of Obesity Using Machine Learning
Brief Title: Machine Learning for Reclassification of Obesity
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The Third People's Hospital of Chengdu (Other); Shanghai East Hospital (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Shen Qu, Clinical Professor and Principal Investigator, Shanghai 10th People's Hospital
Other Study IDs: Obesity Reclassification
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Obesity
Keywords: Obesity; Machine learning; Metabolic classification; Clustering; Bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Adiposity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- NW: normal weight control
- MHO: metabolic healthy obesity
  Interventions: Diagnostic Test: AI classification of patients with obesity
- LMO: hypometabolic obesity
  Interventions: Diagnostic Test: AI classification of patients with obesity
- HMO-U: hypermetabolic obesity with hyperuricemia
  Interventions: Diagnostic Test: AI classification of patients with obesity
- HMO-I: hypermetabolic obesity with hyperinsulinemia
  Interventions: Diagnostic Test: AI classification of patients with obesity

INTERVENTIONS:
Diagnostic Test: AI classification of patients with obesity — Computational modeling techniques will be used for the precise reclassification of obesity into four subgroups, several variables according to the clinical experience and the modeling results will be selected for the cluster analysis.
  Groups: HMO-I; HMO-U; LMO; MHO

SUMMARY:
The goal of this study is to employ or develop computational modeling techniques for the precise reclassification of obesity into subgroups. Clinical features, risks of noncommunicable diseases, as well as weight loss effects of bariatric surgery will also be studied and compared within the subgroups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with overweight/obesity
2. Patients with normal weight as controls

Exclusion Criteria:

1. had ever been performed with a bariatric surgery before the study's first visit is scheduled;
2. had taken exogenous insulin, medication that affects glucose metabolism, or uric acid drugs currently;
3. being diagnosed with type 1 diabetes, secondary diabetes, hereditary disease, or severe disease (e.g. malignant tumor, heart failure, liver failure, etc.);
4. in gestation of lactation;
5. did not have the complete data for model;
6. for normal-weight controls, patients with diabetes or hyperuricemia were excluded.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with overweight/obesity.
Sampling Method: Probability Sample
Enrollment: 2495 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Metabolic classification of patients with obesity using machine learning | baseline

SECONDARY OUTCOMES:
Metabolic features in patients of different subgroups | baseline
Risks for noncommunicable disease in patients of different subgroups | baseline
Effect of bariatric surgery in patients of different subgroups | 1 year after bariatric surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin Z, Feng W, Liu Y, Ma C, Arefan D, Zhou D, Cheng X, Yu J, Gao L, Du L, You H, Zhu J, Zhu D, Wu S, Qu S. Machine Learning to Identify Metabolic Subtypes of Obesity: A Multi-Center Study. Front Endocrinol (Lausanne). 2021 Jul 14;12:713592. doi: 10.3389/fendo.2021.713592. eCollection 2021. PMID 34335479